# Interprofessional Mindfulness Practices Advancing Cancer Teamwork (IMPACT) Research Study

NCT06423183 6/17/2024

# University of Wisconsin - Madison Research Participant Information and Consent Form

**Study Title:** Interprofessional Mindfulness Practices Advancing Cancer Teamwork (IMPACT)

Research Study

Principal Investigator: Lee Wilke, MD (Phone: (608) 266-6400) (Email:

wilke@surgery.wisc.edu)

# Description of the research

You are invited to participate in a research study about how a mindfulness-based team training can improve well-being and team resilience in interprofessional oncology teams. You have been asked to participate because you are a healthcare professional working in oncology care.

The purpose of the research is to understand how we can improve well-being and teamwork in caring for oncology patients.

This study will include healthcare professionals in oncology teams, including clinic nurses, nurse managers, medical assistants, social workers, technicians, nutritionists, pharmacists patient navigators, advanced practice providers, and/or physicians.

This research will be conducted at UW-Madison and UW Health Carbone Cancer Center.

# What will my participation involve?

If you decide to participate in this research, you will be asked to participate in a mindfulness team training that involves 4 sessions over 4 months. The first session will be in-person, and the following sessions will be virtual. The sessions will be recorded so you can view them at a later date. You will be asked to complete online questionnaires before the first session, after the last session, and 3-months after the training. These questionnaires will take 5-10 minutes. You will also be asked to participate in a 30-minute focus group, if you are willing, after the training ends to get your feedback on the training.

Your participation will last approximately 50-60 minutes per session and will require 4 sessions. The training sessions and questionnaires will require 3.5-4 hours in total.

#### **Recording information**

Video and audio tapes will be made of your participation.

Recordings of the sessions will be shared with all study participants on a secure UW drive for viewing during the study. This may include audio or video of you if you participate in discussion during these sessions. If you decide to participate in the focus group, audio recording of that session will be recorded and transcribed.

The tapes/recordings will be kept until the end of the study before they are destroyed.

# Are there any risks to me?

Potential risks for study participants are minimal, and include the following:

You may experience psychological discomfort or distress when completing questionnaire measures. The questionnaires will not assess mental health diseases such as depression or suicidality. During the training, you may be asked to engage in mindfulness-based practices that may involve experiencing unpleasant internal experiences (e.g., worry, repetitive thoughts). There is a minimal risk of loss of confidentiality for research participants in this study.

# Are there any benefits to me?

Participants may find personal benefit from the team resilience training, as it provides tools and practices that can enhance mindfulness skills, social connection, self-awareness, and teamwork. It may improve well-being for individual participants.

### Will I be compensated for my participation?

If you participate in this study and fill out all questionnaires, you will receive a \$10 gift card. A randomly selected participant will be drawn at the end of the study. That participant's clinic or team will receive a \$300 gift card for a team lunch.

# How will my confidentiality be protected?

This study is confidential. Neither your name or any other identifiable information will be published.

Participant data will be handled with the highest degree of confidentiality and discretion. Only approved study personnel will have access to the data.

If you participate in this study, we would like to be able to quote you directly without using your name. If you agree to allow us to quote you in publications, please initial the statement at the bottom of this form.

# Whom should I contact if I have questions?

You may ask any questions about the research at any time. If you have questions, concerns, or complaints, or think that participating in the research has hurt you, talk to the research team or contact the Principal Investigator Lee Wilke, MD at (608) 266-6400.

If you have concerns about your rights as a research participant or have complaints about the research study or study team, call the confidential research compliance line at 1-833-652-2506. UW Staff not part of the study team will work with you to address concerns and assist in resolving any complaints.

If you decide not to participate or to withdraw from the study, you may do so without penalty.

Your signature indicates that you have read this consent form, had an opportunity to ask any questions about your participation in this research and voluntarily consent to participate. You will receive a copy of this form for your records.

| Name of t | he Participant (please print): |
|---|---|
| Signature: | |
| Date: | |
| | I give my permission to be quoted directly in publications without my name. |